CLINICAL TRIAL: NCT01335997
Title: A Phase III Multicenter, Double-Blind, Crossover Design Study to Evaluate Lipid-Altering Efficacy and Safety of 1 g/10 mg Extended-Release Niacin/Laropiprant/Simvastatin Combination Tablets in Patients With Primary Hypercholesterolemia or Mixed Dyslipidemia
Brief Title: Efficacy and Safety of Extended-Release Niacin/ Laropiprant/Simvastatin Tablets in Participants With Hypercholesterolemia or Mixed Dyslipidemia (MK-0524B-143)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0524B-143; 2011-001007-12 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Results first posted 2016-06-21 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Low-density lipoprotein; LDL; High-density lipoprotein; HDL; Niacin; Lipid modifying therapy; Cholesterol; High cholesterol; Triglycerides
MeSH Terms: conditions — Hypercholesterolemia | interventions — MK-0524; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERN/LRPT/SIM → ERN/LRPT+SIM (Experimental): Weeks 0-4 (Period 1): Participants will take ERN/LRPT/SIM 1 g/10 mg and SIM-matching placebo tablets daily; Weeks 5-12 (Period 2): Participants will be advanced to ERN/LRPT/SIM 2 g/20 mg and SIM-matching placebo tablets daily; Weeks 13-20 (Period III): Participants will crossover to ERN/LRPT 2 g + SIM 20 mg coadministration treatment.
  Interventions: Drug: ER niacin/laropiprant (ERN/LRPT); Drug: ER niacin/laropiprant/simvastatin (ERN/LRPT/SIM); Drug: Simvastatin (SIM); Drug: Placebo Run-In; Drug: SIM-matching placebo
- ERN/LRPT+SIM → ERN/LRPT/SIM (Active Comparator): Weeks 0-4 (Period I): Participants will take ERN/LRPT co-administered with SIM (ERN/LRPT 1g + SIM 10 mg tablets) daily; Weeks 5-12 (Period II): Participants will be advanced to ERN/LRPT 2 g + SIM 20 mg daily; Weeks 13-20 (Period III): Participants will crossover to the ERN/LRPT/SIM 2 g/20 mg combination treatment and SIM-matching placebo tablets.
  Interventions: Drug: ER niacin/laropiprant (ERN/LRPT); Drug: ER niacin/laropiprant/simvastatin (ERN/LRPT/SIM); Drug: Simvastatin (SIM); Drug: Placebo Run-In; Drug: SIM-matching placebo

INTERVENTIONS:
Drug: ER niacin/laropiprant (ERN/LRPT) — ER niacin 1 g/laropiprant 20 mg oral tablet taken once daily
  Other Names: MK-0524B
Drug: ER niacin/laropiprant/simvastatin (ERN/LRPT/SIM) — ER niacin 1 g/laropiprant 20 mg/simvastatin 10 mg oral tablet taken once daily
  Other Names: MK-0524A, Tredaptive™
Drug: Simvastatin (SIM) — Simvastatin 10 mg oral tablet taken once daily
  Other Names: Zocor®
Drug: Placebo Run-In — Placebo matches both ER niacin 1 g/laropiprant 20 mg oral tablet and ER niacin 1 g/laropiprant 20 mg/simvastatin 10 mg oral tablet; placebo is taken once daily
Drug: SIM-matching placebo — Placebo for simvastatin 10 mg oral tablet taken once daily

SUMMARY:
This study is being done to find out if tablets containing extended release (ER) niacin, laropiprant, and simvastatin (ERN/LRPT/SIM) are as effective as tablets containing ER niacin and laropiprant taken with simvastatin tablets (ERN/LRPT + SIM) for lowering high cholesterol and high lipid levels in the blood. The primary hypothesis is that ERN/LRPT/SIM 2 g /20 mg is equivalent to ERN/LRPT 2 g coadministered with simvastatin 20 mg in reducing low-density lipoprotein cholestrol (LDL-C).

ELIGIBILITY:
Inclusion criteria:

* Has a history of primary hypercholesterolemia or mixed dyslipidemia and meets LDL-C and triglyceride criteria.
* Is high risk coronary heart disease (CHD) and has LDL-C ≤190 mg/dL (≤4.91 mmol/L).
* Is not high risk CHD and has LDL-C ≤240 mg/dL (≤6.21 mmol/L).

Exclusion criteria:

* Is pregnant or breast-feeding, or expecting to conceive or donate eggs or sperm during the study.
* Has a history of malignancy within ≤5 years, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Consumes more than 3 alcoholic drinks per day (14 per week).
* Is a high risk CHD patient on lipid modifying therapy (LMT).
* Is on any LMT with equivalent or greater LDL-C-lowering efficacy than simvastatin 40 mg.
* Has Type 1 or Type 2 diabetes mellitus that is poorly controlled, or on statin therapy.
* Currently engages in vigorous exercise or is on an aggressive diet regimen.
* Has uncontrolled endocrine or metabolic disease, uncontrolled gout, kidney or hepatic disease, heart failure, recent peptic ulcer disease, hypersensitivity or allergic reaction to niacin or simvastatin, recent heart attack, stroke or heart surgery.
* Is human immunodeficiency virus (HIV) positive.
* Has taken niacin >50 mg/day, bile-acid sequestrants, 3-hydroxy-3-methylglutaryl-coenzyme A(HMG-CoA) reductase inhibitors, ezetimibe, Cholestin™ [red yeast rice] and other red yeast products within 6 weeks, or fibrates within 8 weeks of randomization visit (Visit 3).

Note: Fish oils, phytosterol margarines and other non-prescribed therapies are allowed provided participant has been on a stable dose for 6 weeks prior to Visit 2 and agrees to remain on this dose for the duration of the study.

* Is currently receiving cyclical hormonal contraceptives or intermittent use of hormone replacement therapies (HRTs) (e.g., estradiol, medroxyprogesterone, progesterone). Note: Participants who have been on a stable dose of non-cyclical HRT or hormonal contraceptive for greater than 6 weeks prior to Visit 1 are eligible if they agree to remain on the same regimen for the duration of the study.
* Is taking prohibited medications such as systemic corticosteroids, potent inhibitors of Cytochrome P450 3A4 (CYP3A4), cyclosporine, danazol, or fusidic acid.
* Consumes >1 quart of grapefruit juice/day.
* Requires warfarin treatment and has not been on a stable dose with a stable International Normalized Ratio (INR) for at least 6 weeks prior to Visit 1.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synsopsi Link — http://www.merck.com/clinical-trials/study.html?id=0524B-143&kw=0524B-143&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sequence 1 (randomized) = 577; Sequence 2 (randomized) = 562
Groups:
- ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1): Study drug was administered as extended-release niacin/laropiprant/simvastatin combination (ERN/LRPT/SIM) during Period I and II for 12 weeks and extended-release niacin/laropiprant (ERN/LRPT) + simvastatin (SIM) during Period III for 8 weeks.
- ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2): Study drug was co-administered as extended-release niacin/laropiprant (ERN/LRPT) + simvastatin (SIM) (ERN/LRPT + SIM) during Periods I and II for 12 weeks and extended-release niacin/laropiprant/simvastatin combination (ERN/LRPT/SIM) during Period III for 8 weeks.
Period: Period I and II
Arm/Group | ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1) | ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2)
Started | 577 | 562
Completed | 84 | 83
Not Completed | 493 | 479
Not completed — Adverse Event | 63 | 43
Not completed — Noncompliance with Study Drug | 1 | 1
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Study Terminated by Sponsor | 406 | 415
Not completed — Protocol Violation | 9 | 10
Not completed — Physician Decision | 2 | 1
Period: Period III
Arm/Group | ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1) | ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2)
Started | 84 | 83
Completed | 6 | 4
Not Completed | 78 | 79
Not completed — Adverse Event | 0 | 2
Not completed — Study Terminated by Sponsor | 77 | 76
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1) | ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2) | Total
Number analyzed (Participants) | 577 | 562 | 1139
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (10.44) | 56.4 (10.44) | 56.3 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345 | 332 | 677
  Male | 232 | 230 | 462

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) Blood Levels
Description: Due to study termination caused by the decision to stop the development of the combination tablet, sufficient data were not available to perform the planned efficacy analysis, which is based on the cross-over data collected in period II and III.
Time Frame: Baseline and Week 12 and Week 20
Population: Completers Population - participants that completed the study, have respective endpoint data available at baseline, end of period II and end of period III and were not off study drug more than 3 days prior to their period II and period III observations.
Arm/Group | ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1) | ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C) Blood Levels
Description: as for outcome 1
Time Frame: Baseline and Week 12 and Week 20
Population: as for outcome 1
Arm/Group | ERN/LRPT/SIM → ERN/LRPT+SIM (Sequence 1) | ERN/LRPT+SIM → ERN/LRPT/SIM (Sequence 2)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 22 weeks, including 14 days after last dose of study drug (non-serious adverse events up to 20 weeks and serious adverse events up to 22 weeks)
Description: The All Participants as Treated (APaT) population consisted of all randomized participants who received at least one (1) dose of study treatment post-randomization. Participants were included in the treatment sequences corresponding to the study treatment they actually received.
Groups:
- Seq 1 (Periods I+II): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA: ERN/LRPT/SIMVA 1 g/10 mg for 4 weeks (Period I) followed by ERN/LRPT/SIMVA 2 g/20 mg for 8 weeks (Period II)
- Seq 2 (Periods I+II): ERN/LRPT+SIM → ERN/LRPT/SIM: ERN/LRPT 1 g + SIMVA 10 mg for 4 weeks (Period I) followed by ERN/LRPT 2 g + SIMVA 20 mg for 8 weeks (Period II)
- Seq 1 (Period III): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA: ERN/LRPT 2 g + SIMVA 20 mg for 8 weeks (Period III)
- Seq 2 (Period III): ERN/LRPT+SIM → ERN/LRPT/SIM: ERN/LRPT/SIMVA 2 g/20 mg for 8 weeks (Period III)
Arm/Group | Seq 1 (Periods I+II): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA | Seq 2 (Periods I+II): ERN/LRPT+SIM → ERN/LRPT/SIM | Seq 1 (Period III): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA | Seq 2 (Period III): ERN/LRPT+SIM → ERN/LRPT/SIM
Serious Adverse Events (participants affected / at risk) | 11/567 | 5/554 | 0/83 | 1/82
Other Adverse Events (participants affected / at risk) | 103/567 | 95/554 | 0/83 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seq 1 (Periods I+II): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA (N=567) | Seq 2 (Periods I+II): ERN/LRPT+SIM → ERN/LRPT/SIM (N=554) | Seq 1 (Period III): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA (N=83) | Seq 2 (Period III): ERN/LRPT+SIM → ERN/LRPT/SIM (N=82)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seq 1 (Periods I+II): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA (N=567) | Seq 2 (Periods I+II): ERN/LRPT+SIM → ERN/LRPT/SIM (N=554) | Seq 1 (Period III): ERN/LRPT/SIMVA → ERN/LRPT+SIMVA (N=83) | Seq 2 (Period III): ERN/LRPT+SIM → ERN/LRPT/SIM (N=82)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (43) | 29 (33) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 78 (90) | 72 (78) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated for business reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.